CLINICAL TRIAL: NCT02726893
Title: A Predictive Model for Inadequate Bowel Preparation Before Colonoscopy: Development and Validation
Status: Completed | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice president of Qilu Hospital, Shandong University
Other Study IDs: 2016SDU-QILU-01
Record Dates: First submitted 2016-03-25; First posted 2016-04-04 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Bowel Cleansing Quality; Predictors; Colonoscopy; Boston Bowel Preparation Scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients undergoing colonoscopy: patients undergoing colonoscopy were observed in terms of the bowel preparation quality which is measured by Boston Bowel Preparation Scale (BBPS).
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention

SUMMARY:
About 30% of patients were reported to suffer inadequate bowel preparation.

DETAILED DESCRIPTION:
Risk factors, such as diabetes, constipation, history of intra-abdominal or pelvic surgery, etc, have been demonstrated to be important predictors for inadequate bowel preparation. The aim of the study is to create and verify a predictive model for inadequate bowel preparation in Chinese.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing colonoscopy.
* patients older than 18 years.

Exclusion Criteria:

* patients referred for emergency colonoscopy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. patients undergoing colonoscopy.
  2. patients older than 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 1504 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
inadequate bowel preparation, defined as a Boston Bowel Preparation Scale (BBPS) score. | 5 months
  inadequate bowel preparation

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China